CLINICAL TRIAL: NCT06384716
Title: Evaluation of the Influence of a Core Muscle Control-Based Rehabilitation Program on Pelvic Floor Function in Patients With Multiple Sclerosis
Brief Title: Evaluation of the Influence of a Core Muscle Control-Based Rehabilitation Program Patients With Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEB
Record Dates: First submitted 2024-04-08; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis; Pelvic Floor Disorders; Incontinence, Urinary
MeSH Terms: conditions — Multiple Sclerosis; Pelvic Floor Disorders; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: This is a randomised clinical trial. The research will be conducted in accordance with the framework of application of the Helsinki declaration (21) and the law on Personal Data Protection and guarantee of digital rights (Organic Law 3/2018) . The design of this project will follow the definition of the standard elements of a clinical trial protocol: SPIRIT declaration
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group 1 (Experimental): The intervention group will come to receive the treatment focused on training the motor control of the CORE. This intervention will consist of two sessions per week in which different levels of intervention will be established:
  1. - First week: Sensitisation and voluntary work of the pelvic floor musculature without increasing the increase in intra-abdominal pressure.
  2. - Second week: Work on respiratory motor control and activation of the pelvic floor.
  3. - Third and fourth week: Motor control work with progressive increase in intra-abdominal pressure.
  4. - Fifth and sixth week: Work on dynamic motor control in dual-task situations.
  5. - Seventh and eighth week: Core motor control work in functional activities.
  Interventions: Other: rehabilitation programme based on motor control of core muscles
- Control group (No Intervention): The control group will be evaluated before and after 8 weeks and will continue with their usual treatment.

INTERVENTIONS:
Other: rehabilitation programme based on motor control of core muscles — The exercises performed during the intervention aim to improve the functionality of MS patients and to assess how this can improve pelvic floor health, quality of life, sexual health and urinary incontinence. A specific exercise programme has been designed and will be carried out by physiotherapists specialised in neurological physiotherapy for this purpose. The ultimate aim of the research is to be able to benefit other MS patients from our findings and to propose specific interventions in these areas. However, it is possible that no direct benefit will be obtained after the intervention. At the end of the research you will be informed, if you wish, about the main results and general conclusions of the study. The study does not pose any risk to your health as it is a non-invasive study and no harmful or deleterious action is incurred for the additional collection of the necessary records.
  Arms: Experimental Group 1

SUMMARY:
Given the structural relationship of the CORE as a whole, in this study we propose an intervention based on the global motor control of all the structures that make up the CORE to assess its effectiveness on urinary incontinence, sexual dysfunction and balance, as well as its relationship with respiratory function. According to our hypothesis, a global intervention could also be taken into account during conventional treatment in the future, helping to prevent genitourinary dysfunctions derived from alterations in motor control.

DETAILED DESCRIPTION:
Main objective:

To establish the effect of core motor control training on pelvic floor functionality in patients with multiple sclerosis.

Specific objective: To assess the effect of core motor control training on urinary incontinence.

* To assess the effect of core motor control training on urinary incontinence in patients with multiple sclerosis.
* To assess the effect of core motor control training on quality of life in patients with multiple sclerosis.
* To assess the effect of core motor control training on sexual dysfunction in patients with multiple sclerosis.
* To assess the effect of core motor control training on balance in patients with multiple sclerosis.
* To test the relationship between respiratory functionality and pelvic floor dysfunctions in patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* - Age between 18 and 70 years.
* Confirmed diagnosis of Multiple Sclerosis based on McDonald criteria, with an evolution time of more than two years (remitting or progressive) (24).
* Multiple Sclerosis Disability Status Scale (EDSS) score between 2 (minimal disability in one of the functional systems), and 7.5 (inability to take more than a few steps. Limited to wheelchair and transfer support. Ability to move the chair, but not all day if the chair is conventional and lacks a motor) (25, 26).
* Stable medical treatment for at least six months prior to surgery (26).
* Absence of cognitive impairment, with ability to understand instructions and score 24 or higher on the Minimental Test (27).
* Urinary incontinence as a consequence of neurological involvement.

Exclusion Criteria:

* - Diagnosis of another neurological disease or musculoskeletal disorder other than MS.
* Diagnosis of any cardiovascular, respiratory, genitourinary, metabolic or other conditions that may interfere with this study.
* Having presented urinary incontinence prior to the diagnosis of MS.
* Have suffered an exacerbation or hospitalisation in the last 3 months before starting the assessment protocol, or during the therapeutic intervention process.
* Have received a course of intravenous or oral steroids 6 months prior to the start of the assessment protocol and within the intervention period of the study duration.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the percentage of initial and final maximum activity of the pelvic floor muscles. | 8 weeks
  EMG
- Differences between the initial and final thickness of the oblique abdominis and transverse oblique muscles by ultrasound. | 8 weeks
  US
- Differences in the assessment of health-related quality of life before and after the intervention measured with the I-QOL questionnaire. | 8 weeks
  IQOL
- Differences in the assessment of female UI before and after intervention using the I-CIQ questionnaire | 8 weeks
  I-CIQ

SECONDARY OUTCOMES:
- Difference in the percentage of initial and final maximum activity of the paravertebral musculature activity. | 8 weeks
  EMG
- Differences between initial and final amplitude of initial and final diaphragmatic excursion by ultrasound. | 8 weeks
  US
- Difference between initial and final FVC/- Differences between the initial and final peak expired volume (FEV1) | 8 weeks
  spirometry
differences between peak expiratory pressure (PEM) and minimum initial and end inspiratory pressure (MIP). | 8 weeks
  PIM/PEM
balance | 8 weeks
  trunk control test and Berg Balance test

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Estrada-Barranco, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Cecilia Estrada Barranco, Madrid, Spain